CLINICAL TRIAL: NCT00584948
Title: Characterization and Treatment of CNS Abnormalities in Premutation Carriers: A Double-Blind Placebo-Controlled Trial of Memantine
Brief Title: Memantine Treatment in Fragile X-Associated Tremor/Ataxia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200715426-1; 1RL1AG032115-01 (NIH)
Record Dates: First submitted 2007-12-22; First posted 2008-01-02 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Fragile X-Associated Tremor/Ataxia Syndrome; Fragile X Premutation Carriers
Keywords: FXTAS, Fragile X Premutation
MeSH Terms: conditions — Fragile X Tremor Ataxia Syndrome | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memantine (Experimental)
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Week 1: Take 5mg tab every morning. Week 2: Take 5mg tab every morning and evening. Week 3: Take 10mg tab in the morning and 5 mg in the evening. Week 4: Take 10 mg tab in the morning and evening, and remain on this dose through the remainder of the study.
  Other Names: Namenda
  Arms: Memantine
Drug: Placebo — Week 1: Take 5mg tab every morning. Week 2: Take 5mg tab every morning and evening. Week 3: Take 10mg tab in the morning and 5 mg in the evening. Week 4: Take 10 mg tab in the morning and evening, and remain on this dose through the remainder of the study.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if memantine is effective in treating symptoms of Fragile X-associated Tremor Ataxia Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Fragile X premutation carrier (CGG repeat 55-200)with neurological symptoms; Clinical FXTAS Stage 1-5

Exclusion Criteria:

* Previous reaction to memantine

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randi J Hagerman, MD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - UC Davis MIND Institute, Sacramento, California
  - University of Colorado Health Sciences Center, Aurora, Colorado

REFERENCES:
- [Derived] Seritan AL, Nguyen DV, Mu Y, Tassone F, Bourgeois JA, Schneider A, Cogswell JB, Cook KR, Leehey MA, Grigsby J, Olichney JM, Adams PE, Legg W, Zhang L, Hagerman PJ, Hagerman RJ. Memantine for fragile X-associated tremor/ataxia syndrome: a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2014 Mar;75(3):264-71. doi: 10.4088/JCP.13m08546. PMID 24345444

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Memantine | Placebo
Started | 47 | 47
Completed | 34 | 36
Not Completed | 13 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine | Placebo | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.7) | 66.3 (7.0) | 65.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 34
  Male | 32 | 28 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 47 | 47 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 46 | 43 | 89
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 47 | 47 | 94

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Executive Functioning as Measured by the Behavioral Dyscontrol Scale II (BDS-II)
Description: The BDS-II is a 9-item, 27-point instrument that measures executive function as the capacity for behavioral and attentional self-regulation. Total score is a sum of the 9 items, with a range of 0-27, in which a higher score indicates a better performance.
Time Frame: One Year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 34 | 36
units on a scale
  Baseline | 17.44 (5.19) | 16.12 (5.43)
  One Year | 15.66 (4.11) | 15.72 (3.93)

2. Primary Outcome: Change From Baseline in Intention Tremor as Measured by the CATSYS Tremor Scale
Description: The CATSYS is a set of computer assisted diagnostic instruments that can measure intention tremor, postural tremor, postural sway, manual coordination and reaction time. The tremor intensity is defined as the root mean square of accelerations, recorded in the 0.9 Hz to 15.0 Hz band during the test period. Unit is measured in m/s2
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: m/s^2
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 34 | 36
m/s^2
  Baseline | 1.31 (1.02) | 1.05 (0.73)
  One Year | 1.77 (1.78) | 1.89 (2.19)

ADVERSE EVENTS:
Arm/Group | Memantine | Placebo
Serious Adverse Events (participants affected / at risk) | 2/47 | 3/47
Other Adverse Events (participants affected / at risk) | 6/47 | 2/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=47) | Placebo (N=47)
Motor Vehicle Accident (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — One participant was badly injured in a motor vehicle accident and withdrew from the study
Lung Cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — One participant was diagnosed with terminal lung cancer and withdrew from the study
Ovarian Cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1) — One participant was diagnosed with ovarian cancer and withdrew from the study
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — One participant was diagnosed with pneumonia and withdrew from the study
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — One participant had acute appendicitis and required an appendectomy, and withdrew from the study
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=47) | Placebo (N=47)
Constipation (Gastrointestinal disorders) | 6 (10) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No